CLINICAL TRIAL: NCT05198167
Title: Efficacy of Hyperoxygenated Fatty Acids Versus Hydrocolloid Dressings in the Prevention of Pressure Ulcers in Critically Ill Prone Patients
Brief Title: Efficacy of HOFA Versus Hydrocolloid Dressings in the Prevention of PUs in Critically Ill Prone Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Leire Maculet García, Registered Nurse, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H.U.P.H.: 77/21
Record Dates: First submitted 2021-12-15; First posted 2022-01-20 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Prone Position; Pressure Ulcer
Keywords: Nursing Care; Fatty acids; Prevention; Complications
MeSH Terms: conditions — Pressure Ulcer | interventions — Bandages, Hydrocolloid

STUDY DESIGN:
Intervention Model Description: * Group A: Application of hyperoxygenated fatty acids.
  * Group B: Protection of pressure areas with hydrocolloid dressing.
Who Masked: Outcomes Assessor
Masking Description: In this type of study, the aim is to guarantee internal validity by minimizing possible biases, which is why it is important to guarantee the randomization process and the measurement of variables with objectivity criteria. This type of clinical trial does not allow masking the person who performs the intervention, nor the person who measures the main outcome variable, since given the type of patient and the specific care required, it is not possible for a professional outside the patient's care to carry out the assessment of the patient. Blinded analysis of the patients will be guaranteed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperoxygenated Fatty Acids (Experimental): Application of hyperoxygenated fatty acids in pressure zones for prevention of prone position pressure ulcers
  Interventions: Other: Hyperoxygenated fatty acids
- Hydrocolloid dressings (Experimental): Protection of pressure areas with hydrocolloid dressings for the prevention of prone pressure ulcers
  Interventions: Other: Hydrocolloid dressings

INTERVENTIONS:
Other: Hyperoxygenated fatty acids — Application of hyperoxygenated fatty acids in pressure zones for prevention of prone position pressure ulcers
  Arms: Hyperoxygenated Fatty Acids
Other: Hydrocolloid dressings — Protection of pressure areas with hydrocolloid dressings for the prevention of prone pressure ulcers
  Arms: Hydrocolloid dressings

SUMMARY:
Introduction: Prone position (PP) treatment as a rescue strategy for patients with acute respiratory distress syndrome (ARDS) is a technique increasingly used in our daily practice and, as a result of the current health situation due to SARS COV-2, has become the treatment of choice for many patients. Many of the associated complications can be considerably reduced with the implementation of standardized procedures and a team trained and specialized in this technique and its subsequent care.

Aim: To evaluate the efficacy of the use of Hyperoxygenated Fatty Acids (HOFA) compared to the use of hydrocolloid dressings (HCD) in the prevention of Pressure ulcers (PUs) occurrence in critically ill patients in prone position.

Methods: A randomized clinical trial will be conducted to compare the occurrence of PUs and other complications in patients undergoing PP in the ICU of the HUPHM. Two care groups will be formed in which HOFA and hydrocolloid dressings will be used, respectively, following a strict care protocol previously established in the unit. In addition, other variables related to medical and nursing treatment that may influence the appearance of PUs and other complications associated with PP will also be analyzed.

Scientific relevance: PUs have a major socioeconomic and quality of life impact on patients. Dressings and topical agents for prevention are widely used, however, it is unclear which treatment is most effective in preventing PUs in the prone patient.

Keywords: Prone Position; Nursing care; Pressure ulcer; Fatty acids; Prevention; Complications.

DETAILED DESCRIPTION:
INTRODUCTION

Acute Respiratory Distress Syndrome (ARDS) is an acute, diffuse inflammatory lung disease that results in increased pulmonary vascular permeability and decreased aerated lung tissue. It is characterized by hypoxemia, decreased compliance, increased intrapulmonary shunt and physiological dead space. It is estimated that 7.2 persons per 100,000 population suffer from this disease, with a mortality of 42.7% among patients admitted to an Intensive Care Unit (ICU).

Multiple studies have shown that Prone position (PP) alters the mechanics and physiology of gas exchange to result in improved oxygenation, especially if used early (first 48 hours) in appropriate patients. However, it´s carries complications, some associated with prolonged decubitus, as the pressure ulcers (PUs) on the pelvis, thorax, knees and face.

Dressings and topical agents intended for the prevention of skin injuries are widely used. However, it is not clear which ones are most effective in preventing PUs in the prone patient. On the other hand, it is important to take into account the great impact that PUs have on the quality of life of patients, the increase in hospitalization times and the high costs involved, so it´s important to focus nursing care on their prevention.

Given the current variability in the interchangeable use of hydrocolloid dressings (HCD) and hyperoxygenated fatty acids (HOFA) in the prevention of PUs in patients admitted to the ICU, and given that there is insufficient scientific evidence to support the use of one method of prevention versus the other when the critical patient is placed on PP, it was considered necessary to carry out a clinical trial to evaluate the efficacy of both methods in reducing the incidence of skin lesions, as well as their severity.

HYPOTHESIS

PUs in Intensive Care Units have been shown to be multicausal, so that there is a great variability in the incidence of these diseases. Lima et al published in 2017 that the incidence ranged from 3.3% to 52.9%. Also, other reviews similarly such as Tayyib et al in 2016 are ofshow great variability in the prevalence of PUs in Intensive Care Units, with a range from 3-26%.

For that reason, when establishing the comparison between HOFA methods and hydrocolloid dressings, it is expected to find a lower incidence with the use of HOFA. The investigation will start from hypothetical incidences, but with the first patients recruited, the hypothesis will be restated based on the first results obtained.

METHODOLOGY

Design: A randomized controlled clinical trial with two comparison groups will be performed:

* Group A: Application of hyperoxygenated fatty acids.
* Group B: Protection of pressure areas with hydrocolloid dressing.

Study period: It started in June 2021 until the sample size is reached.

Subjects and study setting: All the patients admitted to the ICU of the Majadahonda Puerta de Hierro University Hospital (MPHUH) who are prescribed the prone position. The study has been started at MPHUH. However, given the possibility of reducing the number of patients likely to require PP, and given the need to achieve an adequate sample size, discussions have been initiated with other hospitals that might be interested in participating. Thus, the investigators will start from hypothetical incidences have begun to recruit ICUs from other centers to coordinate a multicenter proposal in the near future. In this case, the Ethical Committee for Research would be informed of the extension of centers.

Multicenter proposal: The study has been initiated at MPHUH. However, given the possibility of reducing the number of patients likely to require prone decubitus, and given the need to achieve an adequate sample size, contact has been initiated with other hospitals interested in participating pending approval by their hospitals. Once approved in each center, a multicenter proposal would be considered in the near future.

Randomization: All patients admitted to the ICU who meet the inclusion criteria will be randomized into two groups, according to a randomization list prepared by Care Research Unit from MPHUH before starting the study, using a pseudo-random number generator program (Epidat program version 3.1). The distribution will be revealed by means of opaque, numbered, sealed and correlated envelopes, at the time the study subject is recruited.

Before performing the PP maneuver, regardless of the assigned group, the hygiene and hydration care established by the Unit's protocols will be carried out. Subsequently, the care assigned to each group will be carried out. Once the group is assigned (HOFA or HCD), an infographic will be placed in the box with a summary of care to ensure continuity of care. In the event that more prone sessions are required, the same care assigned at the beginning will be maintained in the following sessions.

Blinding: In this type of study, the aim is to guarantee internal validity by minimizing possible biases, which is why it is important to guarantee the randomization process and the measurement of variables with objective criteria. This type of clinical trial does not allow masking the person who performs the intervention, nor the person who measures the main outcome variable, since given the type of patient and the specific care required, it is not possible for a professional outside the patient's care to carry out the assessment of the patient. Blinded analysis of the patients will be guaranteed.

Study termination criteria: Data collection will end after the last prone position session of each patient, at the patient's discharge from the Intensive Care Unit or due to death.

The impossibility of performing the care, for clinical reasons or reasons unrelated to the research as described in the study and in the protocol, will also mean the end of the study in that patient, considering valid the data collected, if any, in previous sessions that met the established criteria.

The study will remain active in the Unit until the sample size is completed.

Recruitment and conduct of the study: All patients admitted to the MPHUH ICU are eligible for inclusion in the study. Inclusion will take place at the time of the decision to subject the patient to treatment in the prone position. Once the decision has been made, the corresponding care group will be randomly assigned by means of a blinded envelope, initiating such care before performing the maneuver.

PP treatment is carried out in critically ill or very critically ill patients, previously sedated in most cases, so that, in general, it will not be possible to obtain the patient's prior consent. In addition, given the urgency in some cases of this clinical decision and the prohibition of visits due to the current COVID-19 pandemic, it will not be possible in many cases to obtain prior written informed consent (IC) from the family. Whenever possible, an information sheet and informed consent will be provided to the family in person. If it is not possible to obtain the written IC, the ICU staff will contact a member of the research team or the collaborating medical team, who will be in charge of informing and obtaining, as soon as possible, the IC by means of a telephone call to the reference family member. If the family refuses to participate, the patient will be removed from the study for that reason and the pre-established data cannot be collected. In this case, the subject would be treated as lost to follow-up for cause.

Study variables: The main outcome variable will be the occurrence of PU, location, extent and severity. In addition, other patient profile variables, clinical variables, treatment and care, PP-related complications, adverse events related to the use of HOFA or HCD will be analyzed. All the data to be collected at the different moments of assessment are specified in the field notebook.

Data collection A register will be kept in which all patient data will be included and assigned a code (the same code that corresponds to the randomization envelope: 001, 002, 003, etc.). A Data Collection Sheet will be prepared for each patient. Part of the information will be collected in situ at the time of the PP maneuver. The rest of the data will be collected from the electronic medical record in the clinical programs PICIS and SELENE. All this is detailed in the Field Notebook. Data will be collected at the time of patient inclusion in the study, before and after performing the prone position maneuver, and 24 hours after the maneuver, with the corresponding follow-up in the event of complications. This data collection will be repeated each time the patient requires PP during their stay in the ICU.

At the time of inclusion in the study, a sealed envelope containing the infographic corresponding to the assigned group, the field notebook and the informed consent form will be taken. In this way, if the research team is not present at the time, the personnel in charge of performing the maneuver will be able to collect the initial data in real time. The rest of the variables will be collected, always in coded form, by the research team. An initial sheet with general data relating to the patient at the time of inclusion in the study and an activity sheet with data relating to each prone maneuver will be collected. As many activity sheets will be included as prognoses are performed on the patient.

Statistical analysis Analyses will be performed per assigned protocol. Means, medians, standard deviations and ranges of quantitative variables and percentages of qualitative variables will be presented in tabular form. Different analyses will be carried out to compare the outcome variables in the two groups, using the appropriate statistical tests (parametric and non-parametric), depending on the variables and the characteristics of the distribution. Possible losses to follow-up and the reasons will be recorded. Possible adverse effects will be recorded. Mean differences for qualitative measures and relative risks, absolute and relative risk reductions and number needed to treat qualitative variables will be presented. For all outcome variables, 95% confidence intervals will be presented. The level of statistical significance is set at a level below 0.05. Data analysis will be carried out using SPSS and/or STATA statistical software.

WORK PLAN AND SCHEDULE

WORK PLAN The present study was prepared following the development of the internal protocol "Procedure: Prone Maneuver HUPHM-UCI-PR-089-01", approved by the MPHUH Departments of Quality and Nursing Management in December 2020.

PHASE I. PREPARATORY. During the following months, training of MPHUH ICU personnel was carried out by means of on-line sessions to train all professionals in this technique and in the correct performance of prone position care, as established in the new protocol. At the same time, the design and development of the report of the present research project was carried out, approved by the Ethical Committee for Research of the MPHUH on 24/05/2021, making the appropriate modifications. After its approval, a session was held for all the staff in which the project was presented, informing and involving the whole Unit.

PHASE II. INTERVENTION. In May 2021, conversations were initiated with other hospitals with the possibility of joining the current project, pending approval by their respective Ethical Committees for Research. In June 2021, the pilot study began in the MPHUH ICU, with recruitment of 36 patients included in the study to date.

PHASE III. FOLLOW-UP. The subjects included in the study will be followed up, collecting the pertinent information. The final analysis will be carried out: Statistical analysis of the data collected. Scientific dissemination is foreseen through publication of the results in scientific journals and dissemination in specialized congresses.

ELIGIBILITY:
Inclusion Criteria:

All patients in prone position admitted to the HUPHM ICU who agree to be included in the study or, if they are unable to communicate, the consent is authorized by their referring family member.

Exclusion Criteria:

Patients with previous pressure ulcers in the following prone-related locations: shoulders, thorax, genitals, iliac crest, knees, ankles, facial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2021-06-12 (Actual); Primary Completion 2022-06-12 (Estimated); Study Completion 2023-06-12 (Estimated)

PRIMARY OUTCOMES:
Pressure ulcers | 24 hours
  The main outcome variable will be the appearance of pressure ulcers, location, extension and severity

CONTACTS AND LOCATIONS:
Overall Officials: Leire Maculet-García, RN, Principal Investigator — Hospital Universitario Puerta de Hierro
Locations (1):
- Majadahonda Puerta de Hierro University Hospital, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Araujo MS, Santos MMPD, Silva CJA, Menezes RMP, Feijao AR, Medeiros SM. Prone positioning as an emerging tool in the care provided to patients infected with COVID-19: a scoping review. Rev Lat Am Enfermagem. 2021 Jan 8;29:e3397. doi: 10.1590/1518-8345.4732.3397. eCollection 2021. PMID 33439949
- [Background] Why Prone? Why Now? Improving Outcomes for ARDS Patients. Crit Care Nurse. 2019 Oct;39(5):84. doi: 10.4037/ajcc2019878. No abstract available. PMID 31575599
- [Background] Perrillat A, Foletti JM, Lacagne AS, Guyot L, Graillon N. Facial pressure ulcers in COVID-19 patients undergoing prone positioning: How to prevent an underestimated epidemic? J Stomatol Oral Maxillofac Surg. 2020 Sep;121(4):442-444. doi: 10.1016/j.jormas.2020.06.008. Epub 2020 Jun 18. PMID 32565264
- [Background] Tayyib N, Coyer F. Effectiveness of Pressure Ulcer Prevention Strategies for Adult Patients in Intensive Care Units: A Systematic Review. Worldviews Evid Based Nurs. 2016 Dec;13(6):432-444. doi: 10.1111/wvn.12177. Epub 2016 Oct 6. PMID 27712030
- [Background] Lima Serrano M, Gonzalez Mendez MI, Carrasco Cebollero FM, Lima Rodriguez JS. Risk factors for pressure ulcer development in Intensive Care Units: A systematic review. Med Intensiva. 2017 Aug-Sep;41(6):339-346. doi: 10.1016/j.medin.2016.09.003. Epub 2016 Oct 22. English, Spanish. PMID 27780589
- [Background] Tayyib N, Coyer F, Lewis P. Saudi Arabian adult intensive care unit pressure ulcer incidence and risk factors: a prospective cohort study. Int Wound J. 2016 Oct;13(5):912-9. doi: 10.1111/iwj.12406. Epub 2015 Feb 9. PMID 25662591
- See also: López R, Sánchez B, Lorenzo M. Manejo del Síndrome de Distrés Respiratorio Agudo (SDRA). ¿Qué hay de nuevo? Revista Electrónica AnestesiaR. 2020;12(8):3. — https://doi.org/10.30445/rear.v12i8.848